CLINICAL TRIAL: NCT01232998
Title: Emergency Department Patient Satisfaction Survey in the Imam Reza Hospital , Tabriz ,Iran, 2008
Status: Completed | Type: Observational
Sponsor: Tabriz University (Other)
Other Study IDs: 8711
Record Dates: First submitted 2010-11-01; First posted 2010-11-02 (Estimated); Last update posted 2010-11-02 (Estimated); Status verified 2008-04

CONDITIONS: Community Sample
Keywords: Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Patient Satisfaction with nursing care
- satisfaction of waiting time for first time visit
- patient satisfaction

SUMMARY:
The investigators want to survey Emergency Department Patient Satisfaction in the Imam Reza hospital ,Tabriz ,Iran by questionnaire form . Finally the investigators want to improve the quality services in the department based on the research result.

ELIGIBILITY:
Inclusion Criteria:

* all patients admitted to emergency department

Exclusion Criteria:

* patients didn't sign consent form

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: community sample
Sampling Method: Probability Sample
Enrollment: 504 (Actual)
Dates: Start 2008-06

PRIMARY OUTCOMES:
Patient Satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Tabriz University of Medical Sciences, Daneshgah Street,, Tabriz, East Azarbijan, Iran

REFERENCES:
- [Result] Boudreaux ED, Friedman J, Chansky ME, Baumann BM. Emergency department patient satisfaction: examining the role of acuity. Acad Emerg Med. 2004 Feb;11(2):162-8. PMID 14759959